CLINICAL TRIAL: NCT00330486
Title: The Use of Acamprosate in Alcohol-Dependent Individuals With Bipolar Disorder
Brief Title: Open Label Trial of Acamprosate in Bipolar Alcoholics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HR15882; 5K24DA000435-08 (NIH)
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Alcohol Dependence; Bipolar Disorder
Keywords: Acamprosate; Addiction; Alcoholism; Alcohol dependence; Bipolar disorder; Depression; Impulsivity; Mania; Substance abuse
MeSH Terms: conditions — Alcoholism; Bipolar Disorder; Behavior, Addictive; Depression; Impulsive Behavior; Mania; Substance-Related Disorders | interventions — Acamprosate

INTERVENTIONS:
Drug: Acamprosate

SUMMARY:
The purpose of this study is to determine whether acamprosate (Campral) is safe and effective in treating alcohol dependence in individuals with bipolar disorder. All subjects in the study must be currently stabilized on mood-stabilizing medication. Half of the subjects will receive acamprosate in addition to their mood-stabilizing medication; control subjects will be maintained on their mood-stabilizing medication alone. Measures of alcohol use as well as mood stability will be obtained weekly throughout the active phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-65
* Meet DSM-IV criteria for current (past 90 days) alcohol dependence
* Meet DSM-IV criteria for bipolar I or bipolar II disorder
* Currently on a mood stabilizing medication regimen, including the use of lithium, valproic acid, lamotrigine, and/or antipsychotic agent FDA approved to treat bipolar disorder without any dosage adjustments in the past month
* Must be able to remain free from alcohol for at least 3 days prior to medication initiation
* Subjects must be able to adequately provide informed consent and function at an intellectual level sufficient to allow the accurate completion of all assessment instruments
* Subjects must consent to random assignment and be willing to commit to medication treatment and follow-up assessments

Exclusion Criteria:

* Individuals with a primary psychiatric disorder other than bipolar disorder
* Individuals with an uncontrolled neurologic condition that could confound the results of the study
* Individuals with an uncontrolled medical condition that may adversely affect the conduct of this trial or jeopardize the subject's safety
* Participants with creatine clearance less than or equal to half of normal value as indicated by chem. 7 results conducted at screening visit.
* Concomitant use of other psychotropic medications not allowed per the protocol
* Women of childbearing potential who are pregnant, lactating or refuse to use adequate forms of birth control
* Current suicidal or homicidal risk
* Baseline scores of > 35 on the Montgomery Asberg Depression Rating Scale and/or > 25 on the Young Mania Rating Scale

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-04; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Alcohol use as determined by the time-line follow-back instrument

SECONDARY OUTCOMES:
Mood stability as determined by the Montgomery-Asberg Depression Rating Scale and the Young Mania Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Bryan K. Tolliver, M.D., Ph.D., Principal Investigator — Division of Clinical Neuroscience, Department of Psychiatry, Medical University of South Carolina; Kathleen T. Brady, M.D., Ph.D., Study Director — Division of Clinical Neuroscience, Department of Psychiatry, Medical University of South Carolina
Locations (1):
- Institute of Psychiatry, Medical University of South Carolina, Charleston, South Carolina, United States